CLINICAL TRIAL: NCT01937520
Title: Acupuncture for Reduction of Inflammation in Thyroid and Parathyroid Surgery: Randomized, Prospective Double Blind Pilot Clinical Trial
Brief Title: Acupuncture for Reduction of Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012002417
Record Dates: First submitted 2013-04-24; First posted 2013-09-09 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Thyroid or Parathyroid Surgery
Keywords: acupuncture; inflammation; thyroid; parathyroid
MeSH Terms: conditions — Thyroid Diseases; Inflammation | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental): acupuncture will be administered after induction for a period of 30 minutes, followed by a 30 minute rest period and then resumption of acupuncture for 30 minutes.
  Interventions: Device: acupuncture
- device (Placebo Comparator): no acupuncture will be done on this group of subjects
  Interventions: Device: no acupuncture

INTERVENTIONS:
Device: acupuncture — One half of subjects will receive a standardized acupuncture regiment
  Arms: acupuncture
Device: no acupuncture — placebo
  Arms: device

SUMMARY:
This study is being done because the investigators wish to study ways to improve recovery after surgery. Injury, including surgical injury, causes inflammation. Inflammation is the body's attempt to protect itself and to start the healing process. Some surgical complications are related to the body's natural inflammatory response. Although mainly a healing response, inflammation can also have side effects which delay recovery. The investigators wish to determine the effect of acupuncture on post-operative surgical pain. An increase in pain after surgery can cause distress for patients. Acupuncture is an alternative medicine methodology originating in China that treats patients by manipulating thin, solid needles that have been inserted into acupuncture points in the skin. Acupuncture has been used for the reduction of pain. The investigators would like to see if acupuncture during surgery can provide a lower level of pain, reduced pain medication requirement, and a lower incidence of nausea and vomiting.

DETAILED DESCRIPTION:
Acupuncture has traditionally been used in Asia and is increasingly popular in Western countries to treat a variety of conditions (1). In recent years, acupuncture is widely used to assist in improving pain and inflammatory diseases (2). However, the mechanisms associated with these treatments that influence the immune system are not yet understood.

Cytokines like interleukin-1β (IL-1β), tumor necrosis factor-α (TNF-α), and interleukin-6 (IL-6) are proposed to be proximal mediators in the early stages of inflammation. They modulate many of the early inflammatory response that is induced by tissue injury, infection, or an immune stimulus (3, 4). Although the response is a critical first line of defense against pathogens, when the inflammatory reaction is uncontrolled, it can cause more damage to the host than the initial stimulus. TNF-α is a pro-inflammatory cytokine that is very effective in local and systemic inflammations (5). In addition, TNF-α increases the production of other inflammatory cytokines such as IL-1β, IL-6, and interleukin-18 (IL-18) during the inflammatory process. Therefore, it initially brings infections under control, produces coagulation in the damaged tissue, and stimulates tissue improvement. An excessive increase of TNF-α level causes an extreme immune reaction and contributes to the development of atherosclerosis, shock, endotoxemia, and chronic inflammatory diseases such as rheumatoid arthritis, ankylosing spondylitis, and inflammatory bowel disease (5-7). Yim and colleagues reported a decrease in increased serum TNF-α, IL-6, and interferon gamma levels by arthritis as a result of electroacupuncture treatment (9). In a rat model for ulcerative colitis, acupuncture inhibited the expression of IL-1β and IL-6 (10). It has been reported that acupuncture significantly reduces complete Freund's adjuvant-induced hind paw edema and mouse air pouch inflammation (11, 12). Acupuncture could also improve immune dysfunction after surgical stress both in human and animals (13, 14).

Some cytokines are pro-inflammatory, but others are anti-inflammatory (3). The anti-inflammatory interleukins comprise interleukine-4 (IL-4) and interleukine-10 (IL-10) and these are considered as mediating the down-regulation of immune-inflammatory conditions. Acupuncture for treatment of the ulcerative colitis rats is possibly related with the decrease of IL-1β, a pro-inflammatory cytokine, and the increase of IL-4, an anti-inflammatory cytokine (15).

Therefore, it is reasonable to expect that the protective action of acupuncture is exerted by the modulation of pro- and anti-inflammatory cytokines. The restoration of balance between pro- and anti-inflammatory cytokines by acupuncture gives into the mechanisms underlying the immune-modulation effect of acupuncture.

Inflammation is associated with pain hypersensitivity that is produced by the release of inflammatory mediators. The pro-inflammatory cytokines play an essential role in pain sensitization (16). The peripheral effects of these cytokines on sensitizing nociceptors have been well documented (16). Post-operative surgical pain can cause significant physiologic and psychologic distress for patients. An increase in pain duration and intensity after surgery can contribute to a variety of complications, including delayed ambulation, pulmonary and thromboembolic complications, increased length of hospital stay, and generalized distress and anxiety. Effective post-surgical pain relief requires a multidisciplinary effort and influences patients' satisfaction with care and successful outcomes (17). Acupuncture has been used for a long time for the reduction of pain. In light of these factors, the use of acupuncture that may allow a reduction in the dosage of conventional analgesics is highly valuable because it can lower the incidence of possible adverse effects. Several trials have demonstrated that patients receiving acupuncture prior to surgery have a lower level of pain, reduced opioid requirement, a lower incidence of post-operative nausea and vomiting, and lower sympatho-adrenal responses (18). The local release of β-endorphin could be responsible for the analgesic effect. β-endorphin may be interacting with cytokines to reduce pain and acupuncture may amplify the interaction between β-endorphin and cytokines.

The investigators will ask patients undergoing thyroid and parathyroid surgery to determine how acupuncture restores a balance of pro- and anti-inflammatory cytokines to reduce pain and inflammation before, during, and after surgery. The effect of acupuncture on post-surgical pain will be evaluated.

Protocol A prospective randomized, double-blinded (patient and data collector), study of 30 patients undergoing thyroid or parathyroid surgery under general anesthesia, will be conducted to compare the effects of acupuncture on the levels of circulating cytokines between acupuncture group and control group. The control group is to receive the same anesthetic and surgical techniques without the acupuncture.

The principal investigator will use the Large intestine 4 (LI-4), the Large intestine 11 (LI-11), and the Stomach 36 (ST-36) acupuncture points (acupoints). LI-4 and LI-11 acupoints lie on the Large intestine meridian (pathway). The Large intestine meridian runs through the frontal neck region including the thyroid. LI-4 point is located in the middle of the 2nd metacarpal bone on the radial side and LI-11 point is located at the lateral end of the transverse cubital crease. Acupuncture on these two acupoints showed increased immune-modulatory effects including cytotoxicity of leukocytes (19, 20). ST-36 point is located on the outside of the anterior crest of the tibia and just below the knee. This point is the most commonly used to reduce general body pain (21). The acupuncture procedures will be performed by an anesthesiologist licensed to do so.

After cleaning the skin with alcohol swabs, an acupuncture needle (30 Gauge, 0.30X30 millimeter, Mac Spring Handle Needle, Korea) will be swiftly inserted approximately 5-10 mm deep bilaterally at both LI-4 and LI-11 acupoints of each arm and at ST-36 acupoint of each leg. Electroacupuncture (EA) will be delivered by a stimulator (Digital Electronic Acupunctoscope 4-C, Model AWQ-104L™ Hong Kong, Dist by Lhasa Medical, Weymouth, MA) via electrodes from the stimulator at 10 Hz frequency with the electrical current of continuous wave. This setting showed significant anti-hyperalgesic effects in a rat inflammation model (22, 23) and also inhibited the up-regulation of IL-1β and its messenger Ribonucleic acid (mRNA) compared to the sham control in a rat model of bone cancer pain (24). EA is a particularly therapeutic method in which a small electrical charge is applied to acupuncture needles inserted at the acupoints. EA has the advantage of combining the stimulation of both needles and electricity compared to manual acupuncture alone, and may potentiate the effect of the acupuncture treatment along the meridians. One end of electrode will be attached to the acupuncture needle handle at LI-4 acupoint, and another end will be attached to the acupuncture needle handle at LI-11acupoint bilaterally. For EA on ST-36, one end of electrode will be attached at the right side ST-36 acupoint and another end will be attached at the left side ST-36 acupoint. A symmetrical biphasic wave will be delivered to the electrodes so that the electrode will be alternately positive and negative and the bilateral LI-4, LI-11, and ST-36 acupoints will be stimulated alternately. Mild muscle twitching will be observed.

The investigator will stimulate the acupoints as follows:

1. EA will be performed for 30 min (a time that is similar to that used in clinical practice).
2. EA will stop after 30 min of the treatment, but leave the needles on the acupoints.
3. Subsequently, EA will be re-initiated for an additional 30 min.

This advanced EA technique showed more increased nitric oxide production in the second interval of EA than that of the first interval, and reduced blood pressure at the end of the second interval in our preliminarily study (25). In addition, this technique increased transient receptor potential vanilloid type-1 receptor immunoreactivity in the acupoints compared to that of non-acupoints (26). The advanced EA treatment will be started just before the beginning of surgery.

At the conclusion of the surgical procedure, the acupuncture needles will be removed. The subjects will be awakened and after meeting the criteria for extubation will be transferred to the Post Anesthesia Care Unit (PACU).

Blood Samples A second intravenous line will be placed in the other arm after the induction of anesthesia and prior to surgical incision to collect blood samples. 15 ml of blood will be collected at three time points: (1) preinduction, (2) just after the advanced EA treatment (3) after arrival in PACU and prior to additional medication administration (approximately 120 minutes post preinduction sample). These specimens will be placed into vacutainer tubes with no anti-coagulant. Blood will be drawn with a syringe attached directly to the angiocatheter which has been placed intravenously. To prevent hemolysis, blood will be transferred without a needle, to a vacutainer whose top has been removed. The vacutainer top will be replaced and specimens labeled with study name, subject's study ID number, sample number, and dated. Bloods from the first two time points will be kept refrigerated until the final sample is obtained postoperatively. Blood samples will be transported to the Institute for Complementary and Alternative Medicine/School of Health Related Professions Interprofessional Health Research Laboratory within the Department of Clinical Lab Sciences (G level, Bergen Building, 65 Bergen St., Newark). They will be centrifuged, serum removed, aliquoted, and stored at -80C until analysis.

Laboratory Analysis Samples will be analyzed for levels of cortisol, C-reactive proteins, and cytokines interleukin (IL)-1α, IL-1β, IL-1ra, IL-2, IL-6, IL-8, IL-10, and TNF-α, by appropriate methods, including ELISA or multiplex fluorescent bead technology. All samples will be run in duplicate on with plates and reagents of the same lot. In addition we will test Adrenocorticotropic hormone (ACTH), glucose and insulin to evaluate the response of the stress. Any samples varying greater than 15% between duplicates will be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Not currently pregnant or beast feeding
2. American Society of Anesthesiologists physical status of 1, 2, 3 as determined by your anesthesiologist
3. Patients have a working telephone

Exclusion Criteria:

1. Uncontrolled high blood pressure (systolic > 180 mm Hg (millimeters of mercury), diastolic>110 mm Hg
2. Heart block >than first degree
3. Pacemaker
4. Cardiac muscle is at risk for injury
5. not English speaking
6. Acupuncture within the last 30 days
7. If you have taken ibuprofen, advil aleve, motrin or aspirin with 5 days of the scheduled surgery.
8. Prior history of drug or alcohol dependence
9. If you are unable to feed, dress or bathe yourself
10. If your breathing tube is not removed prior to leaving the operating room.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Grech, MD, Principal Investigator — Rutgers/NJMS; David D Kim, PhD LaC, Principal Investigator — Rutgers/NJMS; Alex Bekker, MD. PhD, Study Chair — Rutgers/NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
data is in results section

REFERENCES:
- [Background] Grech D, Li Z, Morcillo P, Kalyoussef E, Kim DD, Bekker A, Ulloa L. Intraoperative Low-frequency Electroacupuncture under General Anesthesia Improves Postoperative Recovery in a Randomized Trial. J Acupunct Meridian Stud. 2016 Oct;9(5):234-241. doi: 10.1016/j.jams.2016.03.009. Epub 2016 Apr 4. PMID 27776761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in a Same Day Surgery Suite at a academic medical center. The first participant was enrolled on 7/2/13 and last patient enrolled on 7/15/14.
Groups:
- Acupuncture: acupuncture will be administered after anesthesia induction for a period of 30 minutes, followed by a 30 minute rest period and then resumption of acupuncture for 30 minutes.
  acupuncture: One half of subjects will receive a standardized acupuncture regiment
- Sham: no acupuncture will be done on this group of subjects but since they will be under general anesthesia they will not be aware that they are the control group
  no acupuncture: placebo
Period: Overall Study
Arm/Group | Acupuncture | Sham
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients undergoing thyroid or parathyroid surgery under general anesthesia
Groups:
- Sham/Placebo: no acupuncture will be done on this group of subjects. Since they are under general anesthesia they will not realize they are acting as control group
  no acupuncture: placebo
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham/Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Customized [Number; unit: participants]
  <45 years | 6 | 2 | 8
  45 years or older | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Reduced Pain Medication Requirement
Description: analgesia provided in Post Anesthesia Care Unit PACU)
Time Frame: amount of pain medication provided in PACU
Population: All subjects enrolled in study
Measure: Mean (Standard Error); unit: mg of Morphine
Groups:
- Sham/Placebo: no acupuncture will be done on this group of subjects. These subjects will be under general anesthesia and will not be aware that they are in control group.
  no acupuncture: placebo
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 11 | 9
mg of Morphine | 5.43 (1.70) | 7.36 (1.49)

2. Primary Outcome: Visual Acuity Score (VAS)
Description: VAS is a self reported pain scale with a score ranging from 0 to 10. 0= no pain, 10=worst pain possible. Multiple pain sacores were recorded. single value is reported by average
Time Frame: arrival in PACU to 2 hours post operatively
Population: all study participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 11 | 9
units on a scale | 5.36 (0.97) | 6.67 (1.01)

3. Secondary Outcome: (ACTH )Adrenocorticotropic Hormone
Description: All blood samples were collected during general anesthesia, the first prior to surgical incision and electroacupuncture, the second 60 minutes after incision time and at the completion of electroacupuncture, the third after arrival in PACU but before the administration of analgesia. The data below represents female patients only
Time Frame: serum ACTH from baseline/preoperatively,intraoperatively, upon arrival in PACU
Population: females
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
pg/ml
  preoperative | 8.56 (2.60) | 21.32 (7.08)
  intraoperative | 15.26 (12.13) | 21.41 (8.30)
  postoperative | 53.36 (33.84) | 202 (74.37)
  post op<45years | 110 (88.94) | 276.1 (221.9)
  postop>45 years | 19.4 (8.09) | 177.3 (80.96)
  postop<75kg | 15.03 (5.85) | 27.85 (14.35)
  postop>75 kg | 83.48 (68.23) | 376.2 (73.39)

4. Secondary Outcome: Morphine Equivalent
Description: All analgesic treatments were converted to morphine equivalents in milligrams .
Time Frame: PACU to 2 hours post op
Population: females grouped by age (<45 years and 45 years or greater)
Measure: Mean (Standard Error); unit: mg of Morphine
Groups:
- Sham/Placebo: no acupuncture will be done on this group of subjects
  no acupuncture: placebo
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
mg of Morphine
  < 45 years old | 2 (1.16) | 9.75 (2.75)
  > 45 years old | 3.9 (2.52) | 6.68 (1.76)

5. Secondary Outcome: Morphine Equivalent (mg)
Description: morphine equivalent to analyze whether body weight affected the efficacy of electroacupuncture
Time Frame: PACU arrival to 2 hours post op
Population: females with body weight <75 kg and >than 75 kg
Measure: Mean (Standard Error); unit: mg morphine
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
mg morphine
  <75 kg | 3.25 (2.38) | 9.69 (1.48)
  >75 kg | 4.63 (2.63) | 5.5 (2.17)

6. Secondary Outcome: Modified Quality of Recovery Scale
Description: Modified patient self reported scale with 9 questions regarding general well being including ability to eat, free from constant pain, able to manage activities of daily living. 0= worst possible score and 18=best outcome score
Time Frame: Day 1, 2, 3
Population: all females
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
units on a scale
  Day 1 | 14.5 (0.98) | 13.33 (0.85)
  Day 2 | 16 (0.73) | 15.89 (0.75)
  Day 3 | 17.57 (0.3) | 17 (0.33)

7. Secondary Outcome: Cortisol
Description: All blood samples were collected during general anesthesia, the first prior to surgical incision and electroacupuncture, the second 60 minutes after incision time and at the completion of electroacupuncture, the third after arrival in PACU but before the administration of analgesia.
Time Frame: prior to surgical incision, 1 hour following incision, after arrival in PACU
Population: females
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
ng/ml
  preoperative | 173.6 (83.3) | 155.2 (40.37)
  intraoperative | 103.1 (19.93) | 145.2 (26.85)
  postoperative | 267.4 (89.33) | 394.4 (104.6)
  postoperative<45 years | 375.6 (229.1) | 480 (302.1)
  postoperative>45 years | 202.4 (61.55) | 365.8 (116.9)
  postoperative<75 kg | 252.1 (88.76) | 170.7 (67.28)
  postoperative>75 kg | 296 (180.5) | 618.1 (114.6)

8. Primary Outcome: Morphine Equivalent
Description: equivalent doses of morphine for analgesic relief. All analgesic treatments were converted to morphine equivalents in milligrams.
Time Frame: PACU, day 1 , day 2, day 3
Population: since gender impacts the threshold for analgesic and pain the effects of electroacupuncture on females was analyzed. The same number of females were in both groups but since one subject had preexisting levels of TNF>1ug/ml prior to surgery she was eliminated from the dta base
Measure: Mean (Standard Error); unit: mg morphine
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
mg morphine
  PACU | 3.19 (1.59) | 7.36 (1.49)
  Day 1 | 6.31 (2.14) | 9 (2.44)
  Day 2 | 9.84 (3.44) | 7.42 (2.37)
  Day 3 | 7.93 (3.35) | 5.25 (2.32)

9. Primary Outcome: Pain Levels
Description: Visual Acuity scale 0=no pain 10= worst pain possible
Time Frame: PACU, day 1 , day 2, day 3
Population: female patients self reported pain experience following surgery
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
units on a scale
  PACU | 4.88 (1.29) | 6.67 (1.01)
  Day 1 | 6.67 (1.09) | 5.56 (0.96)
  day2 | 5 (1.09) | 5.93 (0.49)
  day3 | 4.28 (0.95) | 3.33 (0.96)

10. Secondary Outcome: Glucose
Description: the first two blood samples were collected during general anesthesia, the first prior to surgical incision and electroacupuncture, the second 60 minutes after incision time and at the completion of electroacupuncture, the third after arrival in PACU but before the administration of analgesia.
Time Frame: serum glucose from baseline to PACU arrival
Population: females
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
mg/dL
  preoperative | 150.4 (11.36) | 164.4 (10.94)
  intraoperative | 154.3 (8.75) | 187.1 (15.82)
  postoperative | 152.8 (7.76) | 208.1 (13.36)
  post op < 45 years | 154.7 (9.39) | 190 (26)
  post op > 45 years | 151.6 (11.88) | 213.3 (15.93)
  postop <75 kg | 144.3 (7.22) | 210.3 (32.46)
  post op >75 kg | 148.5 (9.06) | 206.4 (2.98)

11. Secondary Outcome: Tumor Necrosis Factor (TNF)
Description: First two blood samples were collected during general anesthesia, first prior to surgical incision and Electro-acupuncture (EA), 2nd 60 minutes after incision and EA, third after arrival in PACU but before administration of analgesia. TNF is a critical pyrogen produced during acute phase of a reaction to trauma.
Time Frame: preoperatively-intraoperatively-postoperatively
Population: female subjects
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
pg/ml
  preoperatively | 1.88 (0.67) | 2.14 (0.63)
  intraoperative | 2.09 (0.62) | 2.25 (0.74)
  postoperative | 1.98 (1.0) | 1.9 (0.7)

12. Secondary Outcome: iNTERLEUKIN (IL-2 and IL-4)
Description: both are IL-2 and IL-4 are critical cytokines regulating the cellular response to induce cellular versus hormone immunity. First two blood samples were collected during general anesthesia: first prior to surgical incision and electroacupuncture, second 60 minutes after incision and electroacupuncture and the 3rd after arrival in PACU but before analgesia.
Time Frame: Preoperatively-intraoperatively-postoperatively
Population: all females
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
pg/ml
  IL-2preoperative | 2.64 (1.53) | 4.26 (3.62)
  IL-2intraoperative | 2.38 (1.3) | 3.4 (2.87)
  IL-2 postoperative | 2.33 (1.31) | 2.77 (2.24)
  IL-4 preoperative | 0.52 (0.15) | 0.59 (0.25)
  IL-4 intraoperative | 0.57 (0.27) | 0.56 (0.28)
  IL-4 postoperative | 0.41 (0.12) | 0.37 (0.1)

13. Secondary Outcome: IL-6
Description: First two blood samples were collected during general anesthesia, first prior to Surgical incision and EA, 2nd 60 minutes after incision and EA and the 3rd after arrival in PACU but before administration of analgesia. IL-6 is a critical inflammatory cytokine produced during the acute phase of reaction to trauma
Time Frame: Preoperatively-intraoperatively-postoperatively
Population: total female results; then females divided into age groups (<45 or >45years) and weights groups (<75kg and >75kg)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
pg/ml
  IL-6 preoperatively | 3.58 (0.92) | 4.65 (0.34)
  IL-6 intraoperatively | 4.98 (1.1) | 4.66 (0.4)
  IL-6 postoperatively | 26.96 (10.35) | 27.45 (7.85)
  IL-6 <45 yrs post op | 23.10 (5.3) | 30.9 (6.9)
  IL-6 >45 yrs postop | 29.28 (16.97) | 26.46 (10.14)
  IL-6 <75 kg postop | 37.15 (28.41) | 16 (3.4)
  IL-6 >75 kg postop | 25.44 (4.47) | 36.61 (12.95)

14. Secondary Outcome: IL-10
Description: IL-10 is an anti-inflammatory cytokine marker. First two blood samples were collected during general anesthesia, first prior to surgical incision and EA, 2nd 60 minutes following incision and EA, and the third after arrival in PACU but before administration of analgesia.
Time Frame: Preoperatively-intraoperatively-postoperatively
Population: total females; then those grouped by age (<45years and>45 years) and weight (<75 Kg and >75kg)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
pg/ml
  IL-10 preoperatively | 5.35 (0.93) | 6.0 (0.8)
  IL_10 intraoperative | 7.28 (1.62) | 7.81 (2.22)
  IL-10 postoperative | 16.15 (9.4) | 16.14 (4.07)
  IL-10 <45 yrs postop | 40.23 (13.64) | 13.64 (10.07)
  IL-10 >45 postop | 7.7 (1.19) | 16.86 (4.8)
  IL-10 <75kg postop | 8.6 (1.6) | 10.7 (4.46)
  IL-10>75kg postop | 32.18 (26.58) | 20.47 (6.1)

15. Secondary Outcome: TGFB1
Description: TGFB1 is a pleiotropic factor regulating the immune system and healing. First two blood samples drawn under general anesthesia, first prior to surgical incision and EA, the 2nd 60 minutes after incision and EA, third after arrival in PACU but before administration of analgesia.
Time Frame: Preoperatively-intraoperatively-postoperatively
Population: all females; then females by groups age (<45 years and >45 years) and weight (<75kg and >75kg)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
pg/ml
  preoperative | 7.30 (3.5) | 3.26 (1.53)
  intraoperative | 19.5 (6.28) | 9.4 (3.5)
  postoperative | 35.17 (8.8) | 12.9 (2.65)
  <45 yrs post op | 16.76 (11.37) | 4.89 (0.48)
  >45 yrs postop | 46.2 (9.9) | 15.2 (2.8)
  <75 kg postop | 56.76 (13.51) | 13.96 (5.39)
  >75kg postop | 21.3 (9.2) | 12.11 (2.73)

16. Secondary Outcome: Serum Insulin Level
Description: to determine if electroacupuncture reduced hyperglycemia
Time Frame: preoperative and postoperative
Population: female subjects preoperatively and postoperatively
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Acupuncture | Sham/Placebo
Number analyzed (Participants) | 8 | 9
pg/ml
  preoperative | 257.4 (92.8) | 378.1 (95.05)
  postoperative | 311.2 (50.59) | 325.4 (84.46)

ADVERSE EVENTS:
Time Frame: 3 days postoperatively
Arm/Group | Acupuncture | Sham/Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes